CLINICAL TRIAL: NCT01832792
Title: Guided Self-help for Binge Eating
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Oxford Health NHS Foundation Trust (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Purpose: Treatment
Other Study IDs: OxGSH1
Record Dates: First submitted 2013-04-09; First posted 2013-04-16 (Estimated); Last update posted 2017-04-04 (Actual); Status verified 2017-03

CONDITIONS: Bulimia Nervosa; Eating Disorder Not Otherwise Specified; Binge Eating Disorder
MeSH Terms: conditions — Bulimia Nervosa; Binge-Eating Disorder | interventions — Waiting Lists

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Self-help (Experimental): In this condition, participants complete a self-help intervention with the support of a therapist. This lasts 12 weeks.
  Interventions: Other: Face-to-face self-help; Other: E-mail self-help
- Waiting List (Other): One third of participants will be allocated to a treatment waiting list, after which they will be randomised to one of the other two arms.
  Interventions: Other: Waiting List

INTERVENTIONS:
Other: Face-to-face self-help — Participants in this arm will receive face-to-face self-help; that is, self-help with the support of a therapist, attending the clinic in person.
  Arms: Self-help
Other: E-mail self-help — Participants in this arm will receive e-mail self-help; that is, self-help with the support of a therapist, provided via e-mail.
  Arms: Self-help
Other: Waiting List — Waiting list condition - participants assigned to a waiting list (no intervention) condition
  Arms: Waiting List

SUMMARY:
Guided self-help (GSH) is a recommended first-step treatment for bulimia nervosa, binge eating disorder, and atypical variants of these disorders. The current study proposes to investigate the effectiveness of providing GSH either face-to-face or via e-mail, also using a delayed treatment control condition. Symptom outcomes will be assessed, and an estimate of cost-effectiveness made. Results are proposed to be disseminated locally and internationally (through submission to conferences and peer-reviewed journals), and will hopefully inform local service provision.

Please note that we are only able to offer the intervention to individuals who are currently registered with a General Practitioner that is covered by Oxford Health NHS Foundation Trust - this is typically restricted to practices in Oxfordshire, Buckinghamshire, and parts of Wiltshire.

ELIGIBILITY:
Inclusion Criteria:

* Registration with a General Practitioner covered by Oxford Health NHS Foundation Trust (typically: Oxfordshire, Buckinghamshire, parts of Wiltshire)
* Primary diagnosis of an eating disorder with recurrent binge eating (BN, EDNOS [BN-type] or BED)
* Age above 17.5 years (box below requires whole numbers)

Exclusion Criteria:

* A severe eating disorder (e.g., one complicated by medical issues that would not be best managed by a self-help intervention)
* BMI <18.5
* Rapid weight loss (regardless of BMI)
* current excessive drug use
* active and untreated psychosis (the latter two are usually exclusion criteria to the EDS)

Min Age: 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 122 (Actual)
Dates: Start 2013-08; Primary Completion 2017-03 (Actual); Study Completion 2017-03 (Actual)

PRIMARY OUTCOMES:
EDE-Q | Change in symptoms between Assessment, Start-of-treatment (approx. 3 months later), End-of-treatment (approx. 12 weeks after start of treatment), and 6-month follow-up
  The EDE-Q is given as a measure of eating disorder symptoms in a standardised pack of measures, all given at Assessment, Start-of-treatment, End-of-treatment, and 6-month follow-up. "Assessment" concerns the patient's first contact with the Eating Disorders Service. Start-of-treatment will proceed as soon as possible; at present, the waiting list is around 3 months. Treatment lasts 12 weeks, so End-of-treatment measures will be given approximately 12 weeks after start of treatment. There is a 6-month follow-up. Binge eating is the primary outcome measure, with other eating disorder symptoms as secondary measures. Change in these symptoms will be assessed over the course of treatment.

SECONDARY OUTCOMES:
CORE-OM | Change in symptoms between Assessment, Start-of-treatment (approx. 3 months later), End-of-treatment (approx. 12 weeks after start of treatment), and 6-month follow-up
  The CORE-OM is given as a measure of psychological distress in a standardised pack of measures, all given at Assessment, Start-of-treatment, End-of-treatment, and 6-month follow-up. "Assessment" concerns the patient's first contact with the Eating Disorders Service. Start-of-treatment will proceed as soon as possible; at present, the waiting list is around 3 months. Treatment lasts 12 weeks, so End-of-treatment measures will be given approximately 12 weeks after start of treatment. There is a 6-month follow-up.
RSES | Change in symptoms between Assessment, Start-of-treatment (approx. 3 months later), End-of-treatment (approx. 12 weeks after start of treatment), and 6-month follow-up
  The RSES is given as a measure of self-esteem in a standardised pack of measures, all given at Assessment, Start-of-treatment, End-of-treatment, and 6-month follow-up. "Assessment" concerns the patient's first contact with the Eating Disorders Service. Start-of-treatment will proceed as soon as possible; at present, the waiting list is around 3 months. Treatment lasts 12 weeks, so End-of-treatment measures will be given approximately 12 weeks after start of treatment. There is a 6-month follow-up.
CIA | Change in symptoms between Assessment, Start-of-treatment (approx. 3 months later), End-of-treatment (approx. 12 weeks after start of treatment), and 6-month follow-up
  The CIA is given as a measure of psychological functioning (quality of life) in a standardised pack of measures, all given at Assessment, Start-of-treatment, End-of-treatment, and 6-month follow-up. "Assessment" concerns the patient's first contact with the Eating Disorders Service. Start-of-treatment will proceed as soon as possible; at present, the waiting list is around 3 months. Treatment lasts 12 weeks, so End-of-treatment measures will be given approximately 12 weeks after start of treatment. There is a 6-month follow-up.
HAq-II | End of Session 3 of treatment (3 weeks into treatment)
  The Helping Alliance Questionnaire is given as a measure of therapeutic alliance after Session 3 of treatment (after 3 weeks from start of treatment) and again at end-of-treatment.
Healthcare Use | Change in healthcare use between Start-of-treatment (approx. 3 months later), End-of-treatment (approx. 12 weeks after start of treatment), and 6-month follow-up
  A measure of healthcare use was developed for the study and is given at Start-of-treatment, End-of-treatment, and 6-month follow-up. Start-of-treatment will proceed as soon as possible after assessment; at present, the waiting list is around 3 months. Treatment lasts 12 weeks, so End-of-treatment measures will be given approximately 12 weeks after start of treatment. There is a 6-month follow-up.

OTHER OUTCOMES:
Therapist Time | After every contact with the patient (approx. weekly), including weekly sessions during treatment (12 weeks)
  Therapists are asked to indicate (to the nearest 5 minutes) how much time they spend doing clinical / administrative tasks for each patient (patient name not included). Although there are no formal guidelines for how therapists report their time, it should accurately record all contact with patients, and thus is suggested to be completed approximately weekly.

CONTACTS AND LOCATIONS:
Overall Officials: Paul E Jenkins, DClinPsychol, Principal Investigator — Oxford Health NHS Foundation Trust
Locations (1):
- Oxford Health NHS Foundation Trust, Oxford, Oxfordshire, United Kingdom

REFERENCES:
- [Derived] Jenkins PE, Luck A, Burrows A, Boughton N. Comparison of face-to-face versus email guided self-help for binge eating: study protocol for a randomised controlled trial. Trials. 2014 May 22;15:181. doi: 10.1186/1745-6215-15-181. PMID 24886555